CLINICAL TRIAL: NCT01406288
Title: Outbreak of Hemolytic Uremic Syndrome Linked to Escherichia Coli of Serotype O104:H4 in Bordeaux Urban Area, June 2011: Evaluation of Diagnostic, Prognostic and Pathophysiological Data
Brief Title: Outbreak of Hemolytic Uremic Syndrome Linked to Escherichia Coli of Serotype O104:H4
Acronym: SHU O104 CUB
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2011/26
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Hemolytic-uremic Syndrome; Escherichia Coli Infections
Keywords: hemolytic-uremic syndrome; shiga-toxin-producing E. Coli
MeSH Terms: conditions — Hemolytic-Uremic Syndrome; Escherichia coli Infections | interventions — Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HUS epidemy in Bordeaux, E. coli of the O104H4 serotype
  Interventions: Other: HUS standard coverage care (including in ICU)

INTERVENTIONS:
Other: HUS standard coverage care (including in ICU) — HUS standard coverage care : plasmaphereses - eculizumab - Immunoadsorption

SUMMARY:
The Hemolytic Uremic Syndrome (HUS) in its typical form occurs after a food born infection with a shiga-toxin secreting bacteria, usually Escherichia coli of the O157H7 serotype. An outbreak of bloody diarrhea followed by HUS begun after a collective meal with 120 persons on June 8th, 2011 in Bègles, a city of Bordeaux urban area (CUB).

At least 9 patients, 8 adults and 1 child have been involved in this HUS outbreak, E. coli of the O104:H4 serotype being demonstrated in most patients. This outbreak is remarkable by its preponderance in adults and women, its aggressiveness with multiorgan involvement , i.e. the kidneys, brain, liver, pancreas, and skin.

Pathophysiology, prognosis, and treatment of typical HUS are poorly defined, particularly in adults who are usually not involved in typical E. coli O157H7 HUS.

The aim of the present study is to gain knowledge on these different aspects of the HUS, including response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with HUS concomitant to the outbreak linked to E. coli O104:H4

Exclusion Criteria:

* Patient not willing to participate or to sign informed consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: dinner guest to a collective meal on June 8th, 2011 in Bègles, a city of Bordeaux urban area (CUB).
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Improve scientific knowledge on epidemic HUS in the context of an outbreak of E. coli O104:H4 HUS in the town of Bègles, urban area of Bordeaux, France | during patient hospitalization
  This is an observational propspective study in which all data will be collected on all pertinent aspects of disease, including therapeutic regimens.

SECONDARY OUTCOMES:
evaluate efficiency of therapeutic and diagnostic strategies | during patient hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: christian COMBE, MD, Study Director — University Hospital, Bordeaux; Christian COMBE, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service de Néphrologie, transplantation dialyse - Hôpital Pellegrin, Bordeaux, France